CLINICAL TRIAL: NCT04312620
Title: Evaluation of OCT and Visual Field Changes After Vitrectomy and ILM Peeling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Almoatz bellah zohier Mohammed, doctor, Assiut University
Other Study IDs: ILM peeling
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: ILM Peeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evulate changes in VF and OCT after viterctomy associated with ILM peeling.

DETAILED DESCRIPTION:
Macular epiretinal membrane (ERM) is a disorder of the vitreomacular interface characterized by ﬁbrocellular proliferation on the anterior surface of the internal limiting membrane (ILM) of the macula. Pars plana vitrectomy with ERM removal and inner limiting membrane peeling is the standard surgical treatment for an ERM. ILM peeling is performed to eliminate the scaffold for myoﬁbroblast proliferation and any microscopic ERM in order to prevent ERM recurrence. ILM peeling is indicated for other pathologies other than ERM such as, diabetic macular edema, and macular hole. ILM peeling is a traumatic procedure that may have many effects on the underlying inner retinal layers that may lead to changes in retinal function.

Retinal edema, eccentric scotoma, dissociation of the nerve fiber layer, iatrogenic punctuate chorioretinopathy, and subretinal, retinal, and vitreous hemorrhage are well described secondary to the surgical trauma of peeling in addition to stain toxicity. Investigation of these changes may assist in aiding the development of minimally traumatic techniques for ILM removal .

Evaluation of functional changes may include visual field and Multifocal electroretinography assessment. Visual field defect after vitrectomy a well known post operative complication usually in eyes that underwent fluid air exchange, the cause of visual field defect remain unclear.

Optical Coherence Tomography (OCT), imaging is done to evaluate inner retinal layers after ILM peeling,High myopic eyes might develop more severe, "scattered" inner retinal defects after ILM peeling.

ELIGIBILITY:
Inclusion Criteria:

1. 1-Idiopathic ERM,
2. Primary full thickness macular hole,
3. Lamellar macular hole, and
4. Vitromacular traction.

Exclusion Criteria:

* 1-Patients with a secondary ERM,

  1. diabetic retinopathy,
  2. venous occlusion,
  3. retinal detachment,
  4. uveitis, and
  5. trauma. 2-Other ocular pathologies that could interfere with the functional results

  <!-- -->

  1. dense cataract ,
  2. glaucoma, and
  3. previous retinal surgery.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients withIdiopathic ERM,Primary full thickness macular hole,Lamellar macular hole, andVitromacular traction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-02-09 (Estimated); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
BCVA | 6 months
  ILM peeling

REFERENCES:
- [Background] Noma H, Funatsu H, Sakata K, Harino S, Mimura T, Hori S. Macular microcirculation in hypertensive patients with and without branch retinal vein occlusion. Acta Ophthalmol. 2009 Sep;87(6):638-42. doi: 10.1111/j.1755-3768.2008.01318.x. Epub 2008 Jul 8. PMID 18631327
- [Result] Higashide T, Ohkubo S, Hangai M, Ito Y, Shimada N, Ohno-Matsui K, Terasaki H, Sugiyama K, Chew P, Li KK, Yoshimura N. Influence of Clinical Factors and Magnification Correction on Normal Thickness Profiles of Macular Retinal Layers Using Optical Coherence Tomography. PLoS One. 2016 Jan 27;11(1):e0147782. doi: 10.1371/journal.pone.0147782. eCollection 2016. PMID 26814541